CLINICAL TRIAL: NCT01559194
Title: A Randomized Comparison of a Low Fat or Low Carbohydrate Dietary Pattern for Weight Loss and Impact on Biomarkers Associated With Breast Cancer Risk in Overweight and Obese Premenopausal Women: Lifestyle Eating and Fitness
Brief Title: Low Fat Versus Protein Sparing Diet for Weight Loss & Impact on Biomarkers Associated With Breast Cancer Risk
Acronym: LEAF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Principal Investigator, Electra Paskett, Associate Director for Population Sciences, Comprehensive Cancer Center, Ohio State University; Marion N. Rowley Professor of Cancer Research and Director, Division of Cancer Prevention and Control, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LEAF; OSU 0372 (Other: Ohio State University)
Record Dates: First submitted 2012-03-19; First posted 2012-03-21 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Breast Cancer; Weight Loss
MeSH Terms: conditions — Breast Neoplasms; Weight Loss | interventions — Diet, Fat-Restricted; Exercise; Diet, Carbohydrate-Restricted

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low Fat Diet + Exercise (Active Comparator): Subjects were educated about a low fat diet plus exercise and then followed for weight loss. They were also asked to monitor their physical activity by wearing a pedometer and recording the total steps walked every day.
  Interventions: Behavioral: Low Fat Diet plus exercise
- Low Carbohydrate Diet + Exercise (Active Comparator): Subjects were educated about a low carbohydrate diet plus exercise and then followed for weight loss. They were also asked to monitor their physical activity by wearing a pedometer and recording the total steps walked every day.
  Interventions: Behavioral: Low Carbohydrate diet + Exercise

INTERVENTIONS:
Behavioral: Low Fat Diet plus exercise — Low fat diet plus exercise - Subjects were educated about a low fat diet plus exercise and then followed for weight loss. They were also asked to monitor their physical activity by wearing a pedometer and recording the total steps walked every day.
  Arms: Low Fat Diet + Exercise
Behavioral: Low Carbohydrate diet + Exercise — Low carbohydrate diet plus exercise: Subjects were educated about a low carbohydrate diet and then followed for weight loss. They were also asked to monitor their physical activity by wearing a pedometer and recording the total steps walked every day.
  Arms: Low Carbohydrate Diet + Exercise

SUMMARY:
The primary specific aim of this study was to determine if overweight and obese premenopausal women can lose weight and if long term weight loss impacts biomarkers associated with breast cancer risk.

DETAILED DESCRIPTION:
We examined a low carbohydrate diet (40% carbohydrates, 30% protein, 30% fat) versus a low fat diet (60% carbohydrates, 20% protein, 20% fat) to determine the impact of these dietary patterns, combined with exercise, on weight loss, body shape and body composition.

Inclusion Criteria:

* Aged 30 and older
* Premenopausal (may be confirmed by FSH)
* No previous diagnosis of cancer (except non-melanomatous skin cancer)
* Body mass index between 25-34 kg/m2
* Women must be expected to live in the Columbus area for the next 18 months
* All women must present a letter of medical clearance from their primary care physician

Exclusion Criteria:

* Pregnant women or women who plan to become pregnant during the study period will not be enrolled. Women who become pregnant during the intervention will be withdrawn from the study.
* Women who are already participating in a formal weight loss program (such as Weight Watchers) will not be eligible.
* Women with a medical history that precludes adherence to either of the two dietary patterns will also be excluded. This includes a history of renal insufficiency, gluten enteropathy, Crohn's disease or other medical conditions that significantly impact nutritional status or metabolism. Women with either type I or controlled type II diabetes will be eligible to participate in this trial.
* All medical problems must be managed and controlled. Lipid profile, blood glucose, hemoglobin A1c, and blood pressure will be assessed at the screening visit. These results will be reviewed by the study physician. Women who have abnormal values that, at the discretion of the study physician, would benefit from medical management will be referred to a primary care physician prior to considering them for enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 30 and older
* Premenopausal (may be confirmed by FSH)
* No previous diagnosis of cancer (except non-melanomatous skin cancer)
* Body mass index between 25-34 kg/m2
* Women must be expected to live in the Columbus area for the next 18 months.
* All women must present a letter of medical clearance from their primary care physician.

Exclusion Criteria:

* Pregnant women or women who plan to become pregnant during the study period will not be enrolled. Women who become pregnant during the intervention will be withdrawn from the study.
* Women who are already participating in a formal weight loss program (such as Weight Watchers)will not be eligible.
* Women with a medical history that precludes adherence to either of the two dietary patterns will also be excluded. This includes a history of renal insufficiency, gluten enteropathy, Crohn's disease or other medical conditions that significantly impact nutritional status or metabolism. Women with either type I or controlled type II diabetes will be eligible to participate in this trial.
* All medical problems must be managed and controlled. Lipid profile, blood glucose, hemoglobin A1c, and blood pressure will be assessed at the screening visit. These results will be reviewed by the study physician. Women who have abnormal values that, at the discretion of the study physician, would benefit from medical management will be referred to a primary care physician prior to considering them for enrollment.

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2005-05; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Number of women who lose weight when following 1 of 2 different calorie-restricted diets | 18 months

SECONDARY OUTCOMES:
Number of women that long-term weight loss impacted biomarkers (including Insulin-like growth factor (IGF)- 1 and IGFBP-3) associated with breast cancer risk | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Electra D. Paskett, PhD, Principal Investigator — The Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Result] David P, Buckworth J, Pennell ML, Katz ML, DeGraffinreid CR, Paskett ED. A walking intervention for postmenopausal women using mobile phones and Interactive Voice Response. J Telemed Telecare. 2012 Jan;18(1):20-5. doi: 10.1258/jtt.2011.110311. Epub 2011 Nov 3. PMID 22052963
- [Result] Llanos AA, Krok JL, Peng J, Pennell ML, Vitolins MZ, Degraffinreid CR, Paskett ED. Effects of a walking intervention using mobile technology and interactive voice response on serum adipokines among postmenopausal women at increased breast cancer risk. Horm Cancer. 2014 Apr;5(2):98-103. doi: 10.1007/s12672-013-0168-4. Epub 2014 Jan 17. PMID 24435584
- [Derived] Foraker RE, Pennell M, Sprangers P, Vitolins MZ, DeGraffinreid C, Paskett ED. Effect of a low-fat or low-carbohydrate weight-loss diet on markers of cardiovascular risk among premenopausal women: a randomized trial. J Womens Health (Larchmt). 2014 Aug;23(8):675-80. doi: 10.1089/jwh.2013.4638. Epub 2014 Jul 16. PMID 25029619
- [Derived] Llanos AA, Krok JL, Peng J, Pennell ML, Olivo-Marston S, Vitolins MZ, Degraffinreid CR, Paskett ED. Favorable effects of low-fat and low-carbohydrate dietary patterns on serum leptin, but not adiponectin, among overweight and obese premenopausal women: a randomized trial. Springerplus. 2014 Apr 4;3:175. doi: 10.1186/2193-1801-3-175. eCollection 2014. PMID 24790820
- See also: Jamesline — http://cancer.osu.edu